CLINICAL TRIAL: NCT00233727
Title: Safety and Efficacy of Two Screen-and-Treat Approaches for the Prevention of Cervical Cancer
Brief Title: Screen and Treat for Cervical Cancer Prevention
Acronym: SAT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left University
Sponsor: Columbia University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); EngenderHealth (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAB3373; NCT00494000 (obsolete NCT alias)
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; cervical intraepithelial neoplasia; prevention; cryotherapy; HPV testing; cytology
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HPV DNA Testing + Cryosurgery (Active Comparator): Patients will undergo a "Screen and Treat" program utilizing HPV DNA testing of clinician-collected cervical samples, followed by cryosurgery of screen positive women.
  Interventions: Procedure: HPV DNA Testing + Cryosurgery
- VIA + Cryosurgery (Active Comparator): Patients will undergo a "Screen and Treat" program utilizing visual inspection of the cervix with acetic acid (VIA), followed by cryosurgery of screen positive women.
  Interventions: Procedure: VIA + Cryosurgery
- Delayed Evaluation and Treatment (No Intervention): Patients will undergo a similar screening process at entry, but will be randomized to have evaluation and treatment delayed until 6 months after screening.

INTERVENTIONS:
Procedure: HPV DNA Testing + Cryosurgery — Patients will undergo a "Screen and Treat" program utilizing HPV DNA testing of clinician-collected cervical samples, followed by cryosurgery of screen positive women.
  Arms: HPV DNA Testing + Cryosurgery
Procedure: VIA + Cryosurgery — Patients will undergo a "Screen and Treat" program utilizing visual inspection of the cervix with acetic acid (VIA), followed by cryosurgery of screen positive women.
  Arms: VIA + Cryosurgery

SUMMARY:
The study measures the impact of "screen-and-treat" on the prevalence of high-grade cervical intraepithelial neoplasia and cancer (CIN 2+). It is a three-arm, randomized clinical trial comparing two "screen-and-treat" approaches to delayed evaluation as a control. The primary outcome is biopsy-confirmed CIN 2+ at 6 months and significant complications within 6 months of randomization with continued follow-up to detect CIN2+ and other complications up to 36 months post-randomization.

DETAILED DESCRIPTION:
Participants and Clinical Examinations: Unscreened, non-pregnant women 35-65 years of age are enrolled at three closely located clinical sites in Khayelitsha, South Africa. All women provide informed consent, receive counseling for confidential HIV serotesting, a questionnaire, a pregnancy test if not postmenopausal, anonymous HIV serotesting, and a vaginal speculum examination by nurses trained in visual inspection of the cervix with acetic acid (VIA). Cervical specimens are obtained for testing for N. gonorrhea, Chlamydia trachomatis and high-risk types of HPV, and cytology. The cervix is washed with 5% acetic acid and inspected for gross abnormalities or areas of acetowhitening and a 35 mm. photograph taken. Women with significant cervicitis or vulvovaginitis are treated using the syndromic approach. N. gonorrhea or Chlamydia trachomatis positive women receive appropriate therapy. A positive VIA examination is defined as any acetowhite lesion and no attempt is made to differentiate the acetowhitening of metaplasia from CIN. Women with lesions suspicious for cancer, large acetowhite lesions extending over 70% of the cervix or into endocervical canal, and 374 unsuitable for cryotherapy due to severe atrophy, polyps, cervix distorted, cervix not adequately visualized are excluded. These women are referred to colposcopy.

Women are asked to return 2-6 days later for randomization to either: (1) HPV arm in which all HPV DNA positive women receive cryotherapy; (2) VIA arm in which all VIA positive women receive cryotherapy; and (3) a delayed evaluation arm in which women are followed untreated, irrespective of HPV or VIA status. Randomization is done at a patient level using a computer-generated randomization schedule with arm assignments provided to the clinics in sealed envelopes. Cryotherapy is performed by a nurse using N2O and a cryosurgical unit (Wallach Surgical Devices, Orange, CT) using two 3-minute freezes. Cytology results are not available at the time of cryotherapy. Both treated and untreated women are asked to return at 4 weeks for a questionnaire.

At 6 months, colposcopy is done by a physician blinded to arm and clinical information. All acetowhite lesions are biopsied and all have an endocervical curettage. Women with CIN 2+ are treated with LEEP. Examinations in women who became pregnant during the study are postponed until three months post-partum. Blood for anonymous HIV serotesting is obtained. All women who were HPV or VIA-positive at enrollment and a subset who were HPV and VIA-negative (all women enrolled in 2002) are scheduled for repeat colposcopy at 12 months, 24 months and 36 months post-randomization. At these visits, cervical samples are collected and colposcopy and biopsy if indicated is performed.

Laboratory Testing: HPV testing is done using the Hybrid Capture 2 HPV DNA assay and high-risk probe mixture (Digene Corporation, Gaithersburg, MD) at the University of Cape Town. Biopsies are processed at Columbia University and blindly evaluated by a single pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Has a cervix
* Never been screened for cervical cancer
* Not currently pregnant

Exclusion Criteria:

* Has previously had a Pap smear
* Has previously undergone treatment for cervical squamous intraepithelial lesion (SIL)
* Have lesions suspicious for cancer, have large acetowhite lesions extending over 70% of the cervix or into endocervical canal, are unsuitable for cryotherapy because of severe atrophy, polyps, cervix distorted, cervix cannot be adequately visualized
* Is unable to cooperate with study procedures or tolerate the insertion of a speculum

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7123 (Actual)
Dates: Start 2000-01; Primary Completion 2006-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of "Screen and Treat" + Cryosurgery | Up to 12 months from entry into the study
  Cervical Intraepithelial Neoplasia (CIN) Grade 2 or 3 or Cervical Cancer:
  To determine the reduction in prevalence of biopsy-confirmed high-grade SIL (HiSIL) when a "Screen and Treat" program utilizing visual inspection of the cervix with acetic acid (VIA) or HPV DNA followed by immediate cryosurgery of screen positive women is carried out by mid-level practitioners without the use of colposcopy in a low-resource setting.

SECONDARY OUTCOMES:
HIV incidence | 6 months after entry into study
  Comparison of the rates of HIV seroconversion in women treated using cryosurgery with that of demographically similar, untreated women.
Safety of Cryosurgery | Up to 12 months from entry into study
  To determine the complication rate of cryosurgery by evaluating the occurrence of any severe adverse events (e.g. bleeding, infection)associated with the use of cryosurgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lynette Denny, MD, Study Director — University of Cape Town; Thomas C Wright, MD, Principal Investigator — Columbia University
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

REFERENCES:
- [Result] Denny L, Kuhn L, De Souza M, Pollack AE, Dupree W, Wright TC Jr. Screen-and-treat approaches for cervical cancer prevention in low-resource settings: a randomized controlled trial. JAMA. 2005 Nov 2;294(17):2173-81. doi: 10.1001/jama.294.17.2173. PMID 16264158
- [Derived] Kuhn L, Wang C, Tsai WY, Wright TC, Denny L. Efficacy of human papillomavirus-based screen-and-treat for cervical cancer prevention among HIV-infected women. AIDS. 2010 Oct 23;24(16):2553-61. doi: 10.1097/QAD.0b013e32833e163e. PMID 20706107